CLINICAL TRIAL: NCT03781089
Title: Patiromer Efficacy to Reduce Episodic Hyperkalemia in End Stage Renal Disease Patients Treated With Hemodialysis (PEARL-HD)
Brief Title: Patiromer Efficacy to Reduce Episodic Hyperkalemia in End Stage Renal Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00088688
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hyperkalemia; End Stage Renal Disease
Keywords: Hemodialysis
MeSH Terms: conditions — Hyperkalemia; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, open-label trial. Eligible ESRD patients who are on thrice weekly HD schedule will be screened from retrospective review of clinical and laboratory parameters from our clinical practice group. A total of 40 patients (randomized 1:1 study drug: usual care) will be enrolled. Duration of study medication exposure will be 4 weeks. The total duration of study, from enrollment until the end of the washout period will be 7 weeks.
Who Masked: Outcomes Assessor
Masking Description: The study is open-label and therefore the subjects, coordinators and investigators are not blinded to the intervention. Titration of the patiromer will require viewing of the serum potassium values. During the data analysis, however, personnel involved will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patiromer Oral Powder Product (Experimental): Patients randomized to the patiromer arm will initiate on 8.4 g/day (one pack) given once a day with breakfast or lunch (in place of the full dose of phosphate binder), to start at the end of Week 0. The patiromer dose will be titrated based on serum potassium concentrations drawn on HD1 of Weeks 1, 2, and 3. Patiromer will be increased by 8.4 g/day if K ≥ 5.1 meq/L, decreased by 8.4 g/day if K < 4.0 mEq/L, and patiromer will be discontinued if K < 3.5 mEq/L.
  Interventions: Drug: Patiromer Oral Powder Product
- Usual care arm (No Intervention): Patients randomized to the usual care arm will undergo monitoring with laboratory measurements as outlined in the study protocol

INTERVENTIONS:
Drug: Patiromer Oral Powder Product — Patients randomized to the patiromer arm will initiate on 8.4 g/day (one pack) given once a day with breakfast or lunch (in place of the full dose of phosphate binder), to start at the end of Week 0. The patiromer dose will be titrated based on serum potassium concentrations drawn on HD1 of Weeks 1, 2, and 3. Patiromer will be increased by 8.4 g/day if K ≥ 5.1 meq/L, decreased by 8.4 g/day if K < 4.0 mEq/L, and patiromer will be discontinued if K < 3.5 mEq/L. Patients randomized to the usual care arm will undergo monitoring with laboratory measurements as outlined in the study protocol
  Other Names: Valtressa
  Arms: Patiromer Oral Powder Product

SUMMARY:
The purpose of this study is to determine whether once-daily dosing of patiromer will reduce the frequency of hyperkalemic episodes in ESRD (end stage renal disease) study participants who receive conventional hemodialysis (HD). The study objective is to determine if patiromer administered orally once a day with breakfast or lunch will reduce episodes of hyperkalemia in ESRD study participants who receive thrice-weekly HD.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label trial. Eligible ESRD patients who are on thrice weekly HD schedule will be screened from retrospective review of clinical and laboratory parameters from our clinical practice group. A total of 40 study participants (randomized 1:1 study drug: usual care) will be enrolled. Duration of study medication exposure will be 4 weeks. The total duration of study, from enrollment until the end of the washout period will be 7 weeks.

This is a proof of concept study, to determine whether administration of patiromer has the potential to change the risk category for ESRD patients who are on conventional HD schedules. In addition, the study will develop and pilot study procedures that could be implemented in a large-scale clinical trial. By nature of the limited size of the study, the power of the trial will be limited. Reducing serum potassium with the use of low dialysate potassium is actually associated with an increased risk of sudden cardiac death. Furthermore, HD patients already carry a high pill burden, and it is unclear if prescription of an additional oral medication will reduce the frequency of episodic hyperkalemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, age at least 18 years
* ESRD treated with thrice-weekly HD for ≥ 6 months.
* At least two measured pre-dialysis serum [K] ≥ 5.5 mEq/L or one [K] ≥ 6.0 mEq/L noted over the past three months
* Current use of dialysate with potassium concentration ≤ 2 mEq/L
* Typical consumption of at least two meals per day
* Have received customary dietary instruction over prior month
* Considered by the treating physician(s) to be in otherwise stable clinical condition.
* If patient is of childbearing potential, he/she will be willing to avoid pregnancy during the study using an acceptable birth control method.

Exclusion Criteria:

* Not considered by the treating physician(s) to be adherent with recommended dialysis schedule and prescribed medications
* Life expectancy < 3 months
* Dialysis-dependent for less than 6 months
* Non-elective hospitalization in prior 3 months
* Currently prescription of oral potassium supplements
* In the prior 3 months, therapy with oral potassium-lowering medication
* Underlying severe gastrointestinal disorders, including history of ischemic bowel.
* Corrected serum calcium concentration > 10.5 mg/dL in prior three months
* Anticipated kidney transplant within the next 3 months
* Prisoners or others who are involuntarily incarcerated or detained
* Pregnant, breastfeeding, or considering pregnancy.
* Participation in a clinical trial of an experimental treatment within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Middleton, MD, Principal Investigator — Duke University
Locations (1):
- DaVita Dialysis Sites, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Participant level data will not be shared.

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified from a population of individuals who had ESKD and were maintained on thrice-weekly hemodialysis at five outpatient clinics.
Pre-assignment Details: A total of 36 individuals with ESKD were enrolled, and prior to randomization three were withdrawn (one due to severe hyperkalemia, one due to prolonged hospitalization, and one due to failure to obtain a baseline electrocardiogram).
Period: Overall Study
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Started | 17 | 16
Completed | 16 | 15
Not Completed | 1 | 1
Not completed — Constipation | 1 | 0
Not completed — Positive pregnancy test | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.7) | 58.5 (11.1) | 56.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 12 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 14 | 27
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Episodes of Serum Potassium ≥ 5.5 mEq/L
Description: To determine if patiromer administered orally once a day with the mid-day meal will reduce episodes of hyperkalemia in ESRD patients who receive thrice-weekly HemoDiaylsis.
Time Frame: Week 4
Measure: Number; unit: episodes
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 17 | 16
episodes | 13 | 41
Statistical Analysis 1: Comparison: Patiromer Oral Powder Product vs Usual Care Arm; Test type: Other; p = 0.024, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Episodes of Serum Potassium ≥ 5.5 mEq/L Per Participant
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Median (Full Range); unit: episodes per participant
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 16 | 15
episodes per participant | 0 [0 to 3] | 3 [0 to 6]
Statistical Analysis 1: Comparison: Patiromer Oral Powder Product vs Usual Care Arm; Test type: Other; p = 0.024, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Median Daily Dose of Patiromer That Was Given in Treatment Arm
Time Frame: Week 3
Population: Not applicable to the Usual Care arm.
Measure: Median (Standard Deviation); unit: grams/day
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 16 | 0
grams/day | 8.4 (0) |

4. Secondary Outcome: Number of Additional Hemodialysis Treatments Due to Hyperkalemia
Description: To determine the between-group differences in need for additional hemodialysis treatments due to hyperkalemia
Time Frame: 4 weeks
Population: Data not collected. Post-dialysis serum potassium concentration was not measured, therefore unable to determine whether post-treatment hyperkalemia occurred.
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Significant Arrhythmia Events as Detected With Cardiac Monitors at Baseline
Description: Clinically significant cardiac arrhythmias included sustained ventricular tachycardia (VT), ventricular fibrillation, asystolic cardiac arrest, non-sustained VT (≥ 3 beats but < 30 seconds), > 3 second pause), atrial fibrillation (> 30 seconds), premature ventricular contractions > 500/24h or bradycardia (heart rate < 40 for 5 consecutive beats).
Time Frame: Baseline
Population: One participant in Usual Care arm lost the cardiac monitor for week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 16 | 15
Participants
  Premature ventricular contractions | 4 | 2
  Non-sustained VT events | 2 | 2
  Atrial fibrillation | 2 | 2
  Bradycardia events | 0 | 0

6. Secondary Outcome: Number of Participants With Significant Arrhythmia Events as Detected With Cardiac Monitors at Week 4
Description: as for outcome 5
Time Frame: Week 4
Population: One participant in Usual Care arm lost the cardiac monitor for week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 16 | 14
Participants
  Premature ventricular contractions | 2 | 4
  Non-sustained VT events | 3 | 2
  Atrial fibrillation | 2 | 1
  Bradycardia events | 0 | 1

7. Secondary Outcome: Number of Participants Who Completed All Study Visits
Description: To determine feasibility of a large-scale hemodialysis-based trial.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 17 | 16
Participants | 16 | 15

8. Secondary Outcome: Number of Participants With More Than 1000 Premature Ventricular Contractions (PVCs) in 24 Hours
Description: PVCs are irregular contractions that start in the ventricles instead of the atria.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 16 | 15
Participants | 2 | 4

9. Secondary Outcome: Change in Serum Albumin Concentration
Description: To determine the between-group differences in serum albumin concentrations.
Time Frame: 4 weeks
Population: Data not collected due to limited resources.
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Parathyroid Hormone (PTH) Concentration
Description: To determine the between-group differences in PTH concentrations.
Time Frame: 4 weeks
Population: Data not collected due to limited resources.
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Serum Potassium Concentration Two Weeks After Study Drug is Discontinued
Description: To determine the change in serum potassium concentration two weeks after study drug is discontinued
Time Frame: 6 weeks
Population: Data not collected due to limited resources.
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Serum Phosphorus Concentration Two Weeks After Study Drug Has Been Discontinued
Description: To determine the change in serum phosphorus concentration two weeks after study drug has been discontinued
Time Frame: 6 weeks
Population: Data not collected due to limited resources.
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Patiromer Oral Powder Product | Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/17 | 2/16
Other Adverse Events (participants affected / at risk) | 5/17 | 5/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer Oral Powder Product (N=17) | Usual Care Arm (N=16)
Hospitalization for new vascular access (Surgical and medical procedures) | 1 | 0
Thrombosis of arteriovenousfistula (Vascular disorders) | 1 | 0
Arrhythmia (A-Fib) (Cardiac disorders) | 0 | 1
Admitted for dry gangrene and lower extremity wound infection secondary to chronic limb ischemia (Infections and infestations) | 0 | 1
Admitted for Altered Mental Status secondary to cefepime neurotoxicity (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer Oral Powder Product (N=17) | Usual Care Arm (N=16)
Parasthesias (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Pain from permcath placement (Surgical and medical procedures) | 0 | 1
Skin sensitivity to Holter patch (Skin and subcutaneous tissue disorders) | 0 | 1
Bloody stools/diarrhea (Gastrointestinal disorders) | 1 | 0
Boil under left arm (Skin and subcutaneous tissue disorders) | 0 | 1
Scabies (Skin and subcutaneous tissue disorders) | 0 | 1
Hospitalization for new vascular access (Surgical and medical procedures) | 1 | 0
Same day surgery-creation of upper extremity arteriovenous fistula on right arm (Surgical and medical procedures) | 1 | 0
Emergency Room visit due to shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hospitalization for amputation (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03781089/Prot_SAP_000.pdf